CLINICAL TRIAL: NCT05980910
Title: Investigation of Protective and Risk Factors for Quality of Recovery-15 (QoR-15) Score for Patients Undergoing Major Abdominal Surgery- an Multi-center Observational Study
Brief Title: Protective and Risk Factors for QoR-15 for Major Abdominal Surgery
Acronym: Q15MAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 20236103RIND
Record Dates: First submitted 2023-07-21; First posted 2023-08-08 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: Patients Undergoing Major Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major abdominal surgery: Patients undergoing elective major abdominal surgery. The definition of major surgery is the estimated surgery time >= 2 hours.

SUMMARY:
Investigation of post-operative recovery among adult patients receiving major abdominal surgery.

DETAILED DESCRIPTION:
This prospective observational clinical trial aims to evaluate the postoperative recovery status of patients undergoing major abdominal surgery using the Quality of Recovery-15 (QoR-15) questionnaire. The QoR-15 has been highly regarded for its importance and research value in evaluating postoperative recovery in previous studies and has been validated in numerous languages, including Mandarin. Furthermore, the QoR-15 is not only a reflection of the subjective recovery quality but has also been found to be associated with objective indicators such as postoperative complications. Therefore, establishing a database of postoperative QoR-15 variations can play a significant role in improving healthcare quality and serves as a validation indicator for many Enhanced Recovery After Surgery (ERAS) outcomes. The study aims to contribute to improving postoperative care and inform future research in the context of ERAS programs..

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 18years and above.
* (2) Undergoing elective abdominal surgery with an expected surgical time of at least two hours and an expected hospital stay of at least two days.

Exclusion Criteria:

* (1) Age under 18 years. (2) Incapacity to give informed consent. (3) Emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients receiving major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
QoR-15 Scores at postoperative day one and day three | 72 hours
  Measure the QoR-15(Quality of Recovery-15) scores on the first day and third day after major abdominal surgery. The QoR-15 score, derived from a 15-item questionnaire using an 11-point numeric rating scale, ranges from 0 to 150, with higher scores indicating better recovery quality.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hosipital Hsin Chu Branch, Hsinchu
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles PS. More than just morbidity and mortality - quality of recovery and long-term functional recovery after surgery. Anaesthesia. 2020 Jan;75 Suppl 1:e143-e150. doi: 10.1111/anae.14786. PMID 31903564
- [Background] Johnson A, Rice AN, Titch JF, Gupta DK. Identifying Components Necessary for an Enhanced Recovery After Surgery Pathway for Elective Intracranial Surgery: An Improvement Project Using the Quality of Recovery-15 Score. World Neurosurg. 2019 Oct;130:e423-e430. doi: 10.1016/j.wneu.2019.06.108. Epub 2019 Jul 4. PMID 31279110
- [Result] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725